CLINICAL TRIAL: NCT02101346
Title: A Human In Vivo Feeding Study Of The Blood Monocyte Response To Dietary Lipid Intake
Acronym: Lipophage14
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in scientific information obtained resulting in early cessation of protocol.
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: Lipophage-14
Record Dates: First submitted 2014-03-13; First posted 2014-04-02 (Estimated); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — Diet, Fat-Restricted

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy, Round 1 (Experimental): For feeding of 5 different fatty acid meals in order to assess the monocyte response ex vivo Mixed high fat diet Low fat diet Saturated fat diet Monounsaturated fat diet Polyunsaturated fat diet
  Interventions: Dietary Supplement: Mixed High Fat Diet; Dietary Supplement: Saturated fat diet; Dietary Supplement: Monounsaturated fat diet; Dietary Supplement: Polyunsaturated fat diet; Dietary Supplement: Low fat
- Healthy, Round 2 (Experimental): For feeding of 2 different fatty meals, in order to assess the molecular monocyte response and track the fate of fats.
  Saturated fat Triolein 13C
  Interventions: Dietary Supplement: Saturated fat diet; Dietary Supplement: Triolein 13C

INTERVENTIONS:
Dietary Supplement: Mixed High Fat Diet — Healthy, Round 1
  Other Names: HFD
  Arms: Healthy, Round 1
Dietary Supplement: Saturated fat diet — Healthy, Round 1 Healthy, Round 2
  Other Names: SF
Dietary Supplement: Monounsaturated fat diet — Healthy, Round 1
  Other Names: MUFA
  Arms: Healthy, Round 1
Dietary Supplement: Polyunsaturated fat diet — Healthy, Round 1
  Other Names: PUFA
  Arms: Healthy, Round 1
Dietary Supplement: Triolein 13C — Healthy, Round 2
  Other Names: 13C Tr
  Arms: Healthy, Round 2
Dietary Supplement: Low fat — Healthy, Round 1
  Other Names: LF
  Arms: Healthy, Round 1

SUMMARY:
The aim of the present study is to identify the effects of different dietary fats on the body's immune system and how different types of cells respond. There will be two rounds of recruitment in order to satisfy different aims of the study. In the first round, volunteers will be asked to undergo five separate 1-day assessments where you will be given diets in the form of milkshakes differing in amounts of fats. Volunteers recruited for this round will also be given the opportunity to participate in the second round of recruitment and feeding. A second round of recruitment will then take place to complete recruitment, if required. In the second round, volunteers will be asked to undergo two separate 1-day assessments in the form of milkshakes with differing fats, one of which will contain a tracking label added to the food during preparation. This label is in the form of is a 'stable isotope' and safe to consume (used commonly in some medical tests - see below for further information) and will allow the researchers to later find the food particles within blood cells. During these 1-day assessments blood samples will be collected to identify the impact different diets have on the immune system, specifically monocyte cells thought to play an important role in the development of atherosclerosis, a primary cause of cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* healthy men
* aged between 18-65 years (inclusive)
* body mass index of between 18.5-25kg/m2

Exclusion Criteria:

* Female
* Undiagnosed metabolic syndrome (assessed at initial screening)
* Current smokers
* Substance abuse
* Excess alcohol intake
* Significant medical illness including: diabetes, established cardiovascular disease, cancer, gastrointestinal disease (e.g. inflammatory bowel disease or irritable bowel syndrome), kidney, liver or pancreatic disease or autoimmune or inflammatory disease processes.
* Taking regular medications
* Major surgery in last 6 months

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in ICAM-1 expression by monocytes | 3 years
  ICAM-1 is a marker of monocyte activation (inflammation). ICAM-1 expression can be measured using flow cytometry techniques to quantify expression and therefore inflammation.

SECONDARY OUTCOMES:
Intracellular lipid volume | 3 years
  Lipid uptake by monocyte subsets will be measured as a % of cell volume by staining monocytes with Oil-red-O for neutral intracellular lipid. The % of cell volume with lipid will be compared between the 5 interventional arms of the trial (mixed high fat, low fat, saturated fat, monounsaturated fat and polyunsaturated fat meals).
Quantity of dietary fatty acid within postprandial monocytes | 3 years
  The quantity of dietary fat incorporated into a monocyte will be measured through the use of isotope labelled dietary fat that will be tracked using gas chromatography to provide an exact quantity of how much intracellular lipid within the monocyte originated from the dietary intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin J Woollard, BSc MSc PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College, London, United Kingdom